CLINICAL TRIAL: NCT04208360
Title: Clinical Evaluation of AI-aided Auscultation With Automatic Classification of Respiratory System Sounds
Acronym: AIR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: StethoMe (Industry)
Responsible Party: Sponsor
Other Study IDs: StethoMe AIR
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Wheezing; Rhonchi; Crackle; Lung Sound
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: StethoMe stethoscope — Assessing whether use of the StethoMe AI lung sounds analysis software provides clinical benefit by improving the identification of abnormal lung sounds.

SUMMARY:
In the present trial, the StethoMe electronic stethoscope will be used for pulmonary auscultation and recording of lung sounds in the pediatric study population.

DETAILED DESCRIPTION:
Multicenter, international - 2 EU sites (max. 1 in Poland) and a single US site.

Trial centers and investigators will be identified and selected based on their clinical and research experience.

The trial objective is to assess whether use of the StethoMe AI lung sounds analysis software provides clinical benefit by improving the identification of abnormal lung sounds in the categories of wheezes, rhonchi, fine crackles and coarse as compared to pulmonary auscultation by experienced physicians (general practitioners (GPs) and pulmonologists).

The recordings will be used to form a gold standard database of lung sounds as evaluated by an expert, independent panel according to the study protocol. The gold standard database will include approximately equal representation of wheezes, rhonchi, fine crackles and coarse crackles. Moreover, the database will also include recordings without any of the previous descripted pathological sounds. The results of these two analyses, by traditional physician listening and by the StethoMe AI software application, will be assessed for sensitivity and specificity to the gold standard database in detection of the four lung sounds and recordings without defined pathological sounds. The StethoMe AI will be considered to provide clinical benefit if it demonstrates statistically better sensitivity or specificity on any of the four lung sounds as compared to the traditional physician auscultation, together with F1 score analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 months and 18 years old (inclusive) admitted and hospitalized in the pulmonary disease ward (PL and EU).
* Children between 3 months and 18 years old (inclusive) admitted and hospitalized in the pulmonary disease ward or treated in an outpatient clinic (US).
* Informed consent of parents or caregivers, according to local regulations.

Exclusion Criteria:

* Skin/soft tissue disease or local infection at the site of pulmonary auscultation or any other contraindication for the pulmonary auscultation.
* Any concurrent disease or condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the project.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: It is planned to enroll 84 patients into the trial in three trial centers that will be participating in the study. Each center should recruit approximately 33% of study recordings (25-30 patients).
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of wheezes by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of rhonchi by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of coarse crackles by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of fine crackles by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of wheezes by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of rhonchi by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of coarse crackles by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of fine crackles by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of wheezes by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of rhonchi by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of coarse crackles by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of fine crackles by StethoMe AI algorithms in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of wheezes by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of rhonchi by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of coarse crackles by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of fine crackles by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of wheezes by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of rhonchi by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of coarse crackles by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of fine crackles by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of wheezes by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of rhonchi by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of coarse crackles by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of fine crackles by pulmonologists in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of wheezes by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of rhonchi by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of coarse crackles by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Sensitivity for detection of fine crackles by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of wheezes by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of rhonchi by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of coarse crackles by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  Specificity for detection of fine crackles by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of wheezes by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of rhonchi by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of coarse crackles by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  F1 score for detection of fine crackles by general practitioners in comparison to gold standard
Collecting pulmonary auscultation recordings | 24 hours
  - Possibility to perform pulmonary auscultation by physician by using study device with dedicated application, defined as a percentage of enrolled patients in whom the pulmonary auscultation was performed.

IPD SHARING:
Plan to Share IPD: No